CLINICAL TRIAL: NCT05955157
Title: Phase II Randomized Controlled Trial Of Dendritic Cell + Cytokine-Induced Killer Cell Immunotherapy With S-1 Versus S-1 Alone As Maintenance Therapy For Advanced Pancreatic Ductal Adenocarcinoma Patients
Brief Title: Combined S-1 With DC+CIK As Maintenance Therapy For Advanced Pancreatic Ductal Adenocarcinoma
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DECIMATE 3.0
Record Dates: First submitted 2022-12-26; First posted 2023-07-21 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-01

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Advanced Solid Tumor
Keywords: Cell-based Immunotherapy; S-1 combined DC+CIK maintenance treatment; DC+CIK immunotherapy
MeSH Terms: interventions — Immunotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Receiving DC-CIK plus S1 maintenance treatment
  Interventions: Biological: Dendritic cell + Cytokine-induced killer cell (DC+CIK) immunotherapy; Drug: Tegafur Only Product
- Control Group (Active Comparator): Receiving S-1 maintenance treatment alone
  Interventions: Drug: Tegafur Only Product

INTERVENTIONS:
Biological: Dendritic cell + Cytokine-induced killer cell (DC+CIK) immunotherapy — DC+CIK immunotherapy will be administrated with S-1 chemo drug as maintenance treatment for patients with advanced PDAC
  Arms: Treatment Group
Drug: Tegafur Only Product — Tegafur (TS-1) will be administrated alone as maintenance treatment to control group as standard of care

SUMMARY:
The goal of this randomized phase 2 controlled clinical trial is to study safety, efficacy of S-1 combined DC+CIK maintenance therapy compared with S-1 alone in improving clinical benefit rate (CBR) among advanced PDAC patients. The main objectives aim to be achieved through this study are :

1. To evaluate the safety of DC+CIK combined immunotherapy when administered with the chemotherapy S-1 as maintenance therapy following first-line chemotherapy regime to advanced pancreatic ductal adenocarcinoma patients.
2. To demonstrate the superiority of of DC+CIK combined immunotherapy in improving clinical benefit rate (CBR) of advanced pancreatic ductal adenocarcinoma patients when administered with the chemotherapy S-1 as maintenance therapy following first-line chemotherapy regime.
3. To investigate the ability of S-1 combined DC+CIK maintenance therapy in reducing pancreatic ductal adenocarcinoma patients' circulating cancer stem cells (CSCs).

In this study, subjects who achieve at least stable disease or partial response will be randomized in ratio of 1:1 into treatment group: DC-CIK plus S1 (27 patients) and control group: S-1 alone (27 patients). For treatment group, they will be infused with DC first, followed by CIK immune cells on day 1. DC+CIK immunotherapy will be repeated for another 2 times (day 8 and 15) as one cycle. All patients are left to rest for a week (start from day 21) prior to receive another 3 times of infusion (day 28, 35 and 42) if condition allowed. Additional third cycle can be performed on those who tolerate well with no toxicity or respond very well. Patients from treatment group will be assessed for their eligibility to receive booster dose on following conditions: 1) tumour achieves partial response or stable disease and 2) ECOG-PS performance status of 0-2 and 3) doesn't exhibit grade 1 and 2 toxicities to improve tumour control.

Additionally, S-1 will be given twice daily after meals for 2 weeks as first cycle along with DC+CIK. Next second cycle of S-1 will be given after 7-days (1 week) rest. The cycles will be repeated every 21 days until disease progression, unacceptable toxic effects, or withdrawal with consent. Dose of S-1 will be determined according to the body surface area.

Meanwhile, patients from control group will receive S-1 alone as maintenance therapy twice daily after meals for 14 days (2 weeks) as one cycle. The next cycle of S-1 will be given after 7-days rest. The cycles will be repeated every 21 days until disease progression, unacceptable toxic effects, or withdrawal with consent.

DETAILED DESCRIPTION:
This trial is designed as randomized phase 2 controlled clinical trial.

Subjects who fulfill following inclusion criteria will be admitted to this phase 2 trial and will be excluded if they fulfill any one of the exclusion criteria. All patients must have undergone first-line of chemotherapy (either modified FOLFIRINOX or gemcitabine-based) for at least 3 months and achieved at least stable disease. The inclusion criteria are as follow: 1) histologically and cytologically confirmed advanced pancreatic ductal adenocarcinoma according to AJCC (American Joint Committee on Cancer) TNM system; 2) have undergone first-line of chemotherapy (modified FOLFIRINOX or gemcitabine-based) for at least 3 months and achieved at least stable disease; 3) Eastern Cooperative Oncology Group performance status (ECOG-PS) of 0-2; 4) age above 18 ages and 5) life expectancy more than three months. Meanwhile, the exclusion criteria are 1) pregnant and lactating women; 2) concomitant beta-adrenergic drug blockers medication; 3) active infection; 4) current enrollment in another clinical study with an investigational agent and 5) patients who undergo pancreas or metastatic site radiotherapy need to be recovered from the toxicities.

Next, patients who achieve at least stable disease will be checked for peripheral blood mononuclear cells (PBMC) adequacy, hematoprofiling using full blood count (FBC) and their baseline status. This is followed by leukapheresis once all conditions satisfied and met. Apheretic products will be sent to local sponsor-contracted laboratory prior for incubation of patients' immune cells with PDAC antigens under specific medium.

All subjects in this trial have been diagnosed with advanced stage of PDAC and being treated with standard chemo: modified FOLFIRINOX or gemcitabine-based regime for at least 3 months. Once the DC+CIK infusion bags are ready to be manufactured, those who achieve at least stable disease or partial response will be randomized in ratio of 1:1 into treatment group: DC-CIK plus S1 (27 patients) and control group: S-1 alone (27 patients).

For treatment group, DC+CIK infusion bag will be administrated right after 17 days patients discharged. Patients will be infused with DC first, followed by CIK immune cells on day 1. DC+CIK immunotherapy will be repeated for another 2 times (day 8 and 15) as one cycle. All patients are left to rest for a week (start from day 21) prior to receive another 3 times of infusion (day 28, 35 and 42) if condition allowed. DC+CIK immunotherapy will be offered as two cycles for every patient in treatment group.

Additional third cycle can be performed on those who tolerate well with no toxicity or respond very well. Patients from treatment group will be assessed for their eligibility to receive booster dose on following conditions: 1) tumour achieves partial response or stable disease and 2) ECOG-PS performance status of 0-2 and 3) doesn't exhibit grade 1 and 2 toxicities to improve tumour control.

Additionally, S-1 will be given twice daily after meals for 2 weeks as first cycle along with DC+CIK. Next second cycle of S-1 will be given after 7-days (1 week) rest. The cycles will be repeated every 21 days until disease progression, unacceptable toxic effects, or withdrawal with consent. Dose of S-1 will be determined according to the body surface area.

Meanwhile, patients from control group will receive S-1 alone as maintenance therapy twice daily after meals for 14 days (2 weeks) as one cycle. The next cycle of S-1 will be given after 7-days rest. The cycles will be repeated every 21 days until disease progression, unacceptable toxic effects, or withdrawal with consent.

All patients will be followed up for clinical effects of S-1 combined maintenance therapy translated by tumour best overall response towards the treatment, either complete response (CR), partial response (PR), stable disease (SD) outcomes or progression disease (PD) and level of prognostic biomarkers. Besides, all patients will undergo baseline CT/MRI scan within 4 weeks of patient randomization and before immunotherapy being initiated. This is followed by reassessment CT/MRI scan at the end of 8th weeks starting from date of first treatment, and after S-1 combined DC+CIK immunotherapy completed. All patients will be followed-up regularly to monitor disease progression using reassessment CT/MRI scan at eight weeks interval until first PD observed (Timeframe = 12 months).

Patients' blood will be taken before maintenance treatment initiated and after maintenance treatment completed to evaluate serum cytokine concentration changes and level of circulating cancer stem cells (CSCs). Furthermore, blood will also be taken after each cycle of DC+CIK immunotherapy completed to evaluate baseline peripheral immune profile. Serum CA19-9 concentrations will be monitored every 4 weeks using blood test after first cycle of DC+CIK treatment completed.

Two endoscopic-ultrasound (EUS) guided biopsy pancreatic specimens (optional) will be collected from treatment group patients before maintenance treatment given and after completion of second cycle DC+CIK immunotherapy to quantify tumour-infiltrating lymphocytes (TILs), apoptotic protein expressed on tumour cells and apoptotic cells.

Finally, patients will be monitored for side effects, toxicities and response toward treatment weekly starting on day 7th onward after initial DC+CIK administration. All dated events occurring any time after informed consent will be obtained until 7 days (for non-serious AEs) or 30 days (for SAEs) after the last day of study participation.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically and cytologically confirmed advanced pancreatic ductal adenocarcinoma according to AJCC (American Joint Committee on Cancer) TNM system;
2. Have undergone first-line of chemotherapy (modified FOLFIRINOX or gemcitabine-based) for at least 3 months and achieved at least stable disease;
3. Eastern Cooperative Oncology Group performance status (ECOG-PS) of 0-2;
4. Age above 18 ages
5. Life expectancy more than three months.

Exclusion Criteria:

1. Pregnant and lactating women
2. Concomitant beta-adrenergic drug blockers medication
3. Active infection
4. Current enrollment in another clinical study with an investigational agent
5. Patients who undergo radiotherapy to pancreas or metastatic site need to be recovered from the toxicities

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events | 3 months
  Safety of patients towards treatment will be evaluated based on number of adverse events (AEs) and serious adverse events (SAEs) reported.
Incidence of treatment-emergent hematologic side effects | 3 months
  Feasibility of experimental treatment will be evaluated based on result of differential complete blood count.

SECONDARY OUTCOMES:
Clinical benefit rate (CBR) - Change from baseline in tumour burden | 12 months
  Tumour best overall response will be evaluated based on baseline CT/MRI scan, conducted within 4 weeks of patient randomizations and before immunotherapy, followed by reassessment CT/MRI scan at the end of 8th weeks after S-1 combined DC+CIK maintenance therapy completed for both treatment and control group using RECIST Guidelines version 1.1
Efficacy of S-1 combined DC+CIK in controlling tumour | 3 months
  Intratumour analysis of tumour-infiltrating lymphocytes
  EUS-biopsy will be consented toward subjects before enroll the trial. Overall, two endoscopic-ultrasound (EUS) guided biopsy pancreatic specimens (optional) will be collected from treatment group patients before maintenance treatment given and after completion of second cycle DC+CIK immunotherapy. The TILs will be stained using immunohistochemistry method before quantified using H-score under bright-field microscope.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Oncology Department, Ummc, Petaling Jaya, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bear AS, Vonderheide RH, O'Hara MH. Challenges and Opportunities for Pancreatic Cancer Immunotherapy. Cancer Cell. 2020 Dec 14;38(6):788-802. doi: 10.1016/j.ccell.2020.08.004. Epub 2020 Sep 17. PMID 32946773
- [Background] Chen L, Zhang X. Primary analysis for clinical efficacy of immunotherapy in patients with pancreatic cancer. Immunotherapy. 2016 Feb;8(2):223-34. doi: 10.2217/imt.15.105. Epub 2015 Nov 13. PMID 26565954
- [Background] Du H, Yang J, Zhang Y. Cytokine-induced killer cell/dendritic cell combined with cytokine-induced killer cell immunotherapy for treating advanced gastrointestinal cancer. BMC Cancer. 2020 Apr 28;20(1):357. doi: 10.1186/s12885-020-06860-y. PMID 32345239
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Foley K, Kim V, Jaffee E, Zheng L. Current progress in immunotherapy for pancreatic cancer. Cancer Lett. 2016 Oct 10;381(1):244-51. doi: 10.1016/j.canlet.2015.12.020. Epub 2015 Dec 23. PMID 26723878
- [Background] Gammaitoni L, Giraudo L, Leuci V, Todorovic M, Mesiano G, Picciotto F, Pisacane A, Zaccagna A, Volpe MG, Gallo S, Caravelli D, Giacone E, Venesio T, Balsamo A, Pignochino Y, Grignani G, Carnevale-Schianca F, Aglietta M, Sangiolo D. Effective activity of cytokine-induced killer cells against autologous metastatic melanoma including cells with stemness features. Clin Cancer Res. 2013 Aug 15;19(16):4347-58. doi: 10.1158/1078-0432.CCR-13-0061. Epub 2013 Jun 21. PMID 23794732
- [Background] Haag GM, Stocker G, Quidde J, Jaeger D, Lordick F. Randomized controlled trial of S-1 maintenance therapy in metastatic esophagogastric cancer - the multinational MATEO study. BMC Cancer. 2017 Jul 31;17(1):509. doi: 10.1186/s12885-017-3497-9. PMID 28760152
- [Background] He W, Huang Z, Zhou S, Huang L, Wang B, Zhu L, Ding Y, Yu YL, Zhang S. The effect of DC+CIK combined therapy on rat liver cancer model and its modulatory effect on immune functions. Eur Rev Med Pharmacol Sci. 2018 Feb;22(3):778-785. doi: 10.26355/eurrev_201802_14312. PMID 29461610
- [Background] Miller KD, Fidler-Benaoudia M, Keegan TH, Hipp HS, Jemal A, Siegel RL. Cancer statistics for adolescents and young adults, 2020. CA Cancer J Clin. 2020 Nov;70(6):443-459. doi: 10.3322/caac.21637. Epub 2020 Sep 17. PMID 32940362
- [Background] Pan CC, Huang ZL, Li W, Zhao M, Zhou QM, Xia JC, Wu PH. Serum alpha-fetoprotein measurement in predicting clinical outcome related to autologous cytokine-induced killer cells in patients with hepatocellular carcinoma undergone minimally invasive therapy. Chin J Cancer. 2010 Jun;29(6):596-602. doi: 10.5732/cjc.009.10580. PMID 20507732
- [Background] Sudo K, Nakamura K, Yamaguchi T. S-1 in the treatment of pancreatic cancer. World J Gastroenterol. 2014 Nov 7;20(41):15110-8. doi: 10.3748/wjg.v20.i41.15110. PMID 25386059
- [Background] Ueno H, Ioka T, Ikeda M, Ohkawa S, Yanagimoto H, Boku N, Fukutomi A, Sugimori K, Baba H, Yamao K, Shimamura T, Sho M, Kitano M, Cheng AL, Mizumoto K, Chen JS, Furuse J, Funakoshi A, Hatori T, Yamaguchi T, Egawa S, Sato A, Ohashi Y, Okusaka T, Tanaka M. Randomized phase III study of gemcitabine plus S-1, S-1 alone, or gemcitabine alone in patients with locally advanced and metastatic pancreatic cancer in Japan and Taiwan: GEST study. J Clin Oncol. 2013 May 1;31(13):1640-8. doi: 10.1200/JCO.2012.43.3680. Epub 2013 Apr 1. PMID 23547081
- [Background] Wang Z, Liu Y, Li R, Shang Y, Zhang Y, Zhao L, Li W, Yang Y, Zhang X, Yang T, Nie C, Han F, Liu Y, Luo S, Gao Q, Song Y. Autologous cytokine-induced killer cell transfusion increases overall survival in advanced pancreatic cancer. J Hematol Oncol. 2016 Feb 3;9:6. doi: 10.1186/s13045-016-0237-6. PMID 26842696
- [Background] Xie Y, Huang L, Chen L, Lin X, Chen L, Zheng Q. Effect of dendritic cell-cytokine-induced killer cells in patients with advanced colorectal cancer combined with first-line treatment. World J Surg Oncol. 2017 Nov 28;15(1):209. doi: 10.1186/s12957-017-1278-1. PMID 29179719
- [Background] Yuan X, Zhang AZ, Ren YL, Wang XL, Jiang CH, Yang L, Liu CX, Liang WH, Pang LJ, Gu WY, Li F, Hu JM. Cytokine-induced killer cells/dendritic cells and cytokine-induced killer cells immunotherapy for the treatment of esophageal cancer: A meta-analysis. Medicine (Baltimore). 2021 Apr 2;100(13):e24519. doi: 10.1097/MD.0000000000024519. PMID 33787569
- [Background] Zhu H, Yi C, Zhao Y, Gou H. Gemcitabine plus S-1 for metastatic pancreatic cancer. Medicine (Baltimore). 2018 Oct;97(41):e12836. doi: 10.1097/MD.0000000000012836. PMID 30313120

DOCUMENTS (1):
  • Informed Consent Form (2023-01-05): https://cdn.clinicaltrials.gov/large-docs/57/NCT05955157/ICF_000.pdf